CLINICAL TRIAL: NCT06086613
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled, Single and Multiple Ascending-Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AGA2115 in Adult Healthy Volunteers
Brief Title: A First-in-Human Study Evaluating AGA2115 in Adult Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Angitia Incorporated Limited (Industry)
Responsible Party: Sponsor
Organization: Angitia Biopharmaceuticals (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ACT22-002
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2023-10

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- AGA2115 (Experimental): In Part A, up to 6 single ascending dose cohorts.
  In Part B, up to 3 multiple ascending dose cohorts.
  Interventions: Drug: AGA2115
- Placebo (Placebo Comparator): Participants will receive matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AGA2115 — In Part A, participants will receive AGA2115 as a single dose administered as a subcutaneous (SC) injection (5 cohorts) or as an intravenous (IV) infusion (1 cohort).
  In Part B, participants will receive AGA2115 in multiple doses administered as a SC injection.
  Arms: AGA2115
Drug: Placebo — In Part A, participants will receive single dose of placebo administered as a SC injection (5 cohorts) or IV infusion (1 cohort).
  In Part B, participants will receive multiple doses of placebo administered as a SC injection.
  Arms: Placebo

SUMMARY:
To understand if AGA2115 is safe and well tolerated in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women ≥18 to ≤65 years old.
* Vitamin D sufficiency (≥20 ng/mL (50 nmol/L) and agree to taking Calcium and Vitamin D supplements during the trial.

Exclusion Criteria:

* History of myocardial infarction or stroke (or other cardiovascular associated event deemed significant by investigator) within 12 months prior to Day 1.
* Malignancy within the last 5 years (basal cell carcinoma and squamous cell carcinoma that have been excised with no recurrence within the last 5 years is allowed).
* Hyper- or hypocalcemia.
* Known sensitivity to mammalian-derived drug preparations and/or any biologics.
* Pregnant or breastfeeding or planning to become pregnant (self or partner) at any time during the study.

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2023-10-03 (Actual); Primary Completion 2024-10-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) | Day 1 to up to end of study (approximately 85 days in Part A, approximately 169 days in Part B)
  Clinically significant changes in clinical laboratory tests, vital signs, and 12-lead electrocardiograms (ECGs) will be recorded as TEAEs.

SECONDARY OUTCOMES:
Maximum observed concentration (Cmax) of AGA2115 | Day 1 to up to end of study (approximately 85 days in Part A, approximately 169 days in Part B)
Time to maximum observed concentration (Tmax) of AGA2115 | Day 1 to up to end of study (approximately 85 days in Part A, approximately 169 days in Part B)
Area under the concentration time curve (AUC) of AGA2115 | Day 1 to up to end of study (approximately 85 days in Part A, approximately 169 days in Part B)

CONTACTS AND LOCATIONS:
Overall Officials: Angitia Medical Director, Study Director — Angitia Incorporated Limited
Locations (1):
- Orange County Research Center, Lake Forest, California, United States

IPD SHARING:
Plan to Share IPD: No